CLINICAL TRIAL: NCT01218373
Title: Health Monitoring and sOcial Integration environMEnt for Supporting WidE ExTension of Independent Life at HOME (HOMESWEETHOME)
Brief Title: The Clinical Evaluation of Continuous Assistance Offered to Older People Living Independently.
Acronym: HOMESWEETHOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Him SA (Other)
Collaborators: Ziekenhuis Netwerk Antwerpen (ZNA) (Other); EuroCross (Unknown); Badalona Serveis Assistencials (Other); Department of Health, Generalitat de Catalunya (Other Government); Louth County Council (Unknown); Health Services Executive North Eastern Area (Unknown); TeleMedicina Rizzoli (Unknown); Darco Servizi (Unknown); Azienda USL di Latina (Unknown); University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSH-CLTRPR-01; 250449 (Other Grant/Funding Number: European Commission CIP-ICT PSP-2009-3)
Record Dates: First submitted 2010-10-05; First posted 2010-10-11 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Frailty
Keywords: older people; living independently at home
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group: HOMESWEETHOME services (Active Comparator): Monitoring and alarm handling services. eInclusion services. Domotica services. Daily scheduler. Navigation services. Cognitive training services. Non-technology based services.
  Interventions: Device: HOMESWEETHOME Services
- Control Group: No HOMESWEETHOME services (Placebo Comparator): Normal care.
  Interventions: Device: No HOMESWEETHOME services installed

INTERVENTIONS:
Device: HOMESWEETHOME Services — Monitoring and alarm handling services. eInclusion services. Domotic services. Daily scheduler. Navigation services. Cognitive training services. Non-technology based services.
  Other Names: e.g. DREAMING project devices.
  Arms: Intervention Group: HOMESWEETHOME services
Device: No HOMESWEETHOME services installed — Normal care and healthcare without HOMESWEETHOME services.
  Other Names: no applicable
  Arms: Control Group: No HOMESWEETHOME services

SUMMARY:
The clinical evaluation of the HOMESWEETHOME project sets out to assess the long-term effects of continuous assistance offered by the HOMESWEETHOME services to older people living independently. The trial will test the hypothesis that while providing a level of safety equivalent to or better than that enjoyed in older people"s homes, there is a significant positive effect on the quality of life (QoL) and the duration of independently living of older people.

DETAILED DESCRIPTION:
The HOMESWEETHOME clinical trial is conducted as a multi-centre randomised control trial (RCT), across four pilot sites. The trial design, analysis and reporting follow the "Revised CONSORT - Consolidated Standards of Reporting Trials - Statement" and subsequent additions to the CONSORT statement.

HOMESWEETHOME services are expected to result in an outcome that is superior to usual care alone in reducing deterioration of health related quality of life and function associated with age and chronic disease. This effect will be measured by assessing different outcomes.

The clinical evaluation of the HOMESWEETHOME project sets out to assess the long-term effects of continuous assistance offered by the HOMESWEETHOME services to older people living independently. The trial will test the hypothesis that while providing a level of safety equivalent to or better than that enjoyed in older people"s homes, there is a significant positive effect on the quality of life (QoL) and the duration of independently living of older people.

The study is conducted in four sites within the European Union, these sites will have the number of participants randomised into Intervention Group and Control Group, as follows:

* Belgium - City of Antwerp 30 + 30
* Catalonia - Town of Badalona 15 + 15
* Ireland - North Eastern Region 30 + 30
* Italy - Town of Latina 30 + 30 The main inclusion criteria for participants" entry into the trial will be based on frailty. Frailty is a concept associated with adverse outcomes such as higher morbidity, more hospitalisations and falls, and a lower quality of life. Furthermore, frailty predicts - better than age - the evolution to disability and death. Participants must also be 65 years or over, and living at home. The main reasons for excluding participants will be based on their physical or mental (in)ability to take part.

The primary clinical outcome for the trials will be measured based on the Health Status Questionnaire Short Form 36 (SF-36) (v2).

Secondary outcomes will be measured using Edmonton Frailty Scale (EFS), Comprehensive Geriatric Assessment (CGA), Clinical Global Impression (CGI), and Hospital Anxiety and Depression Scale (HADS). A number of medical events will also be measured.

Measurements will be taken at trial start, trial mid-term, and trial end. Measurements will be entered, anonymously, into a database for analysis of results. The trial population size has been subjected to a statistical power analysis, to ensure statistical significance of project results.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or over.
* Living at home or in the community, i.e. not in a nursing home, acute or sub-acute clinical or care setting.
* Scoring "mildly frail" or "moderately frail" in Edmonton Frail Scale (EFS).

Exclusion Criteria:

* Not willing to participate (e.g. no signing informed consent form).
* Living situation not suitable for independent living (also including long planned durations of absence from home).
* Physically, mentally or otherwise unable to use and / or operate HOMESWEETHOME devices / instruments.
* Unable to administer self-assessment measurements (e.g. monitoring vital signs; questionnaires).
* Significant impairment of language comprehension or expression (e.g. aphasia).
* Active medical illness with a significant shortened life expectancy (< 6 months), based on mortality prognosis2.
* Living without access to ISDN or ADSL service.
* Living with another HOMESWEETHOME participant in the same home.
* Completely dependent on others for the activities of daily living.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2010 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) | measurement will be at trial start (t=0 months)
  Health related QoL as measured with Health Status Questionnaire Short Form 36 (SF-36) (v2).
Quality of life (QoL) | measurement will be at trial midterm (t=15 months)
  Health related QoL as measured with Health Status Questionnaire Short Form 36 (SF-36) (v2).
Quality of life (QoL) | measurement will be at trial end (t=30 months)
  Health related QoL as measured with Health Status Questionnaire Short Form 36 (SF-36) (v2).

SECONDARY OUTCOMES:
Nursing home admission | measurement will be at trial start (t=0months)
  Nursing home admission as assessed from records/equivalent sources
Mortality | continous monitoring during trial duration = 30 months.
  deceasing of participant
Frailty | measurement will be at trial start (t=0 months)
  Frailty as assessed with Edmonton Frailty Scale (EFS)
Geriatric assessment | measurement will be at trial start (t=0 months)
  as assesses with Comprehensive Geriatric Assessment (CGA)
Clinical Global Impression | measurement will be at trial start (t=0 months)
  as assessed with Clinical Global Impression (CGI)
Depression and anxiety | measurement will be at trial start (t=0 months)
  as assessed with Hospital Anxiety and Depression Scale (HADS).
Nursing home admission | measurement will be at trial midterm (t=15 months)
  Nursing home admission as assessed from records/equivalent sources
Nursing home admission | measurement will be at trial end (t=30 months).
  Nursing home admission as assessed from records/equivalent sources
Frailty | measurement will be at trial midterm (t=15 months)
  Frailty as assessed with Edmonton Frailty Scale (EFS)
Frailty | measurement will be at trial end (t=30 months)
  Frailty as assessed with Edmonton Frailty Scale (EFS)
Geriatric assessment | measurement will be at trial midterm (t=15 months)
  as assesses with Comprehensive Geriatric Assessment (CGA)
Geriatric assessment | measurement will be at trial end (t=30 months)
  as assesses with Comprehensive Geriatric Assessment (CGA)
Depression and anxiety | measurement will be at trial midterm (t=15 months)
  as assessed with Hospital Anxiety and Depression Scale (HADS).
Depression and anxiety | measurement will be at trial end (t=30 months)
  as assessed with Hospital Anxiety and Depression Scale (HADS).
Clinical Global Impression | measurement will be at trial midterm (t=15 months)
  as assessed with Clinical Global Impression (CGI)
Clinical Global Impression | measurement will be at trial end (t=30 months)
  as assessed with Clinical Global Impression (CGI)
Number of hospitalisations | measurement will be at trial start (t=0 months)
Number of hospitalizations | measurement will be at trial midterm (t=15 months).
Number of hospitalisations | measurement will be at trial end (t=30 months)
Number of accesses to emergency rooms | measurement will be at trial start (t=0 months)
Number of accesses to emergency rooms | measurement will be at trial midterm (t=15 months).
Number of accesses to emergency rooms | measurement will be at trial end (t=30 months)

CONTACTS AND LOCATIONS:
Overall Officials: Wouter A Keijser, MD, Study Director — Him SA
Locations (4):
- ZNA, Antwerp, Flanders, Belgium
- Netwell Centre, Dublin, Ireland
- Viale P.L. Nervi, Centro Commerciale Latinafiori, Torre Girasoli, 4100 Latina, Latina, Lazio Regon, Italy
- Badalona Serveis Assistencials, Badalona, Catalonia, Spain